CLINICAL TRIAL: NCT02580175
Title: Surgical Evacuation of First Trimester Missed Miscarriage With or Without Use of Transabdominal Ultrasound
Brief Title: Surgical Evacuation of Abortion Under Ultrasonographic Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USEV
Record Dates: First submitted 2015-10-17; First posted 2015-10-20 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Abortion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blinded evacuation (Active Comparator): Ring evacuation was performed in the conventional way without use of ultrasound followed by sharp gentle curettage until complete evacuation
  Interventions: Procedure: Blinded evacuation
- Evacuation under ultrasound guidance (Active Comparator): Ring evacuation was performed under ultrasound guidance followed by sharp gentle curettage until complete evacuation. The surgery was considered complete when the endometrial cavity appeared as a regular echogenic line.
  Interventions: Procedure: Evacuation under ultrasound guidance

INTERVENTIONS:
Procedure: Blinded evacuation — Ring evacuation was performed in the conventional way without use of ultrasound followed by sharp gentle curettage until complete evacuation.
  Arms: Blinded evacuation
Procedure: Evacuation under ultrasound guidance — Ring evacuation was performed under ultrasound guidance followed by sharp gentle curettage until complete evacuation. The surgery was considered complete when the endometrial cavity appeared as a regular echogenic line.
  Arms: Evacuation under ultrasound guidance

SUMMARY:
Abortion is considered the most common cause of fetal demise all over the world. The majority of cases occur in the first trimester. The termination of abortion may be by medical or surgical methods, however; the surgical methods represent the greater part of termination. Therefore, the safety of this procedure is a worldwide public health concern. Many clinical studies have reported the safety of surgical evacuation in the first trimester.

The suction-aspiration or vacuum aspiration is the most common surgical method of induced abortion. This consists of removing the fetus, embryo, placenta, and membranes by suction using a manual syringe or electric pump. However; these techniques always need cervical dilation before aspiration. The menstrual extraction does not require cervical dilation and can be used in very early pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women with non-viable first trimester intrauterine pregnancy
* no contraindication to surgical evacuation under general anesthesia

Exclusion Criteria:

* gestational age more than 13 weeks
* hemodynamically unstable
* suspicion of an ectopic pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Measurement of endometrial thickness by ultrasound (mm) | 1 month

SECONDARY OUTCOMES:
Measurement of blood loss (mL) | 1 month
measurement of operative time (minutes) | 1 month
measurement of Hemoglobin level(g/ml) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt